CLINICAL TRIAL: NCT01737489
Title: Title: "Development and Implementation of Innovative Auditory Training Methods and Verification of These Training Methods"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Annamary (Ann) Peterson, AUDIOLOGIST, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-007641
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Cochlear Implant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LACE ( Listening And Communication Enhancement ) (Active Comparator): use the commercially available auditory training program which is administered by computer as daily lessons.
  Interventions: Behavioral: LACE
- NOOK (Electronic reader) (Active Comparator): will use an electronic reader (NOOK device) to do speech tracking
  Interventions: Behavioral: NOOK
- Control (No Intervention)

INTERVENTIONS:
Behavioral: LACE — commercially available LACE program which is administered by computer as daily lessons. The participants will do this program for one month
  Arms: LACE ( Listening And Communication Enhancement )
Behavioral: NOOK — will use an electronic reader (Barnes and Noble - NOOK device) to do speech tracking.will do this activity for approximately one hour per day for five days out of seven for a total of four weeks. The speech tracking activity will involve reading approximately two books within the one month time frame. The participants will listen to the book while reading an unabridged book in printed form.
  Arms: NOOK (Electronic reader)

SUMMARY:
The purpose of this study is to determine if aural rehabilitation adds measurable benefit and participant satisfaction to a cochlear implant recipient's overall treatment. Also, the study is designed to compare the efficacy of a commercially available aural rehabilitation program (LACE) and an electronic program which takes advantage of a traditional form of auditory training (NOOK) for cochlear implant users.

DETAILED DESCRIPTION:
The primary objective of this study is to determine if aural rehabilitation adds measurable benefit and participant satisfaction to a cochlear implant recipient's overall treatment.

The secondary objective of this study is to compare the efficacy of a commercially available aural rehabilitation program (LACE) and an electronic program which takes advantage of a traditional form of auditory training (NOOK) for cochlear implant users.

ELIGIBILITY:
Criteria for Inclusion:

* Willingness to participate
* Ability to provide informed written consent
* Willingness to follow study protocol
* Eighteen years or older at the time of signing the consent form
* Cochlear implant experience for 12 months or greater
* Spoken English as the first language
* Access to a home computer which meets the minimal requirements to run appropriate program or the ability to use an electronic reader depending on which group the participant is assigned to.
* Reports being comfortable using a computer if in the LACE group

Criteria for Exclusion:

* Unable or unwillingness to sign informed written consent
* Unable or unwillingness to follow study protocol
* Non-English speaking or English as a second language
* No access to a computer if assigned to the LACE study group
* Reports not being comfortable using a computer if assigned to the LACE study group.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Word recognition | baseline to 6 months
  Word recognition will be measured using the Consonant Nucleus Consonant (CNC) Test, a 50 word open set test.
Signal-to-noise ratio | baseline to 6 months
  The signal to noise ratio will be measured using the Bamford-Kowal-Bench (BKB) test.

SECONDARY OUTCOMES:
Percent of speech comprehension | baseline to 6 months
  Percent of speech comprehension will be measured by the AzBio Sentence Lists, which were created at Arizona State University and evaluate speech understanding.

CONTACTS AND LOCATIONS:
Overall Officials: Annamary Peterson, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States